CLINICAL TRIAL: NCT02090790
Title: The Compare the Effect of Peroperative Intravenous Single Dose Dexamethasone and the Addition of Dexamethasone to Femoral Nerve Block on Postoperative Analgesic Consumption Anf Patient Comfort in Unilateral Total Knee Arthroplasty Patients
Brief Title: Comparison of Analgesic Consumption Between Perioperative ıv Dexamethasone and Added to Femoral Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ahmet öner, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/400
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Postoperative Pain
Keywords: dexamethasone; femoral block; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- iv dexamethasone (Active Comparator): perioperative 2ml 8 mg ıv dexamethasone
  Interventions: Drug: iv dexamethasone
- femoral dexamethasone (Active Comparator): femoral block was performed postoperative 30 ml 0,5 % bupivacaine added 2 ml 8 mg dexamethasone
  Interventions: Drug: femoral dexamethasone
- serum physiologic (Placebo Comparator)
  Interventions: Drug: serum physiologic

INTERVENTIONS:
Drug: iv dexamethasone — 2 ml 8 mg iv dexamethasone
  Other Names: decort
  Arms: iv dexamethasone
Drug: femoral dexamethasone — 2ml 8mg dexamethasone administration added 30 ml 0,5 % bupivacain
  Other Names: dekort
  Arms: femoral dexamethasone
Drug: serum physiologic — 2 ml iv serum physiologic
  Arms: serum physiologic

SUMMARY:
the aim of this study was to investigate compare the effect of peroperative intravenous single dose dexamethasone and the addition of dexamethasone to femoral nerve block on postoperative analgesic consumption and patient comfort in unilateral total knee arthroplasty patients

DETAILED DESCRIPTION:
Total knee arthroplasty leads to severe postoperative pain. for postoperative pain control after total knee arthroplasty oral -intramuscular opioids ,patient controlled analgesia intravenous or epidural opioids, single -continuous femoral nerve block involving techniques are used.

Dexamethasone is a glucocorticoid of high potency and frequently used perioperative.Dexamethasone to the local anaesthetic solution administered trough in femoral nerve blocks significantly prolonged the analgesic effect of the local anaesthetics used on this blocks.If the analgesic efficacy of systemic treatment with dexamethasone is similar with the use of perineural wich is the safest way should be preferred for systemic use.

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 age
* knee arthroplasty
* no known allergies to drugs
* ASA 1-2 patients

Exclusion Criteria:

* history of diabetes
* history of chronic pain treatment
* pregnancy
* severe bronchopulmonary disease
* systemic opioid and steroid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | postoperative 2 day

SECONDARY OUTCOMES:
analgesic consumption | postoperative 2 day
  morphine consumption (patient controlled analgesia procedure)

CONTACTS AND LOCATIONS:
Overall Officials: ahmet öner, recident, Principal Investigator — erciyes univercity; gülen güler, prof, Study Director — erciyes univercity
Locations (1):
- Erciyes Univercity Hospital, Kayseri, Turkey (Türkiye)